CLINICAL TRIAL: NCT01232309
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study of the Effects of Chitin-Glucan on Oxidized Low-Density Lipoprotein (LDL)
Brief Title: Effects of Chitin-Glucan on Oxidized Low-Density Lipoprotein (LDL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stratum Nutrition (Industry)
Collaborators: Kitozyme (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KSN-CS-001
Record Dates: First submitted 2010-10-30; First posted 2010-11-02 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Cardiovascular
Keywords: Arterial Health; Fiber; Chitin-glucan; oxidized LDL
MeSH Terms: interventions — carboxymethyl-chitin-glucan; olive extract; Flour

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- High Dose Chitin-Glucan (Active Comparator): Daily oral dose of 4.5 g of chitin-glucan
  Interventions: Dietary Supplement: Chitin-Glucan
- Low Dose Chitin-Glucan (Active Comparator): Daily oral dose of 1.5 g chitin-glucan
  Interventions: Dietary Supplement: Low Dose Chitin-Glucan
- Low Dose Chitin-Glucan + Olive Extract (Experimental): Daily oral dose of 1.5 g chitin-glucan + 135 mg olive extract
  Interventions: Dietary Supplement: Low Dose Chitin-Glucan + Olive Extract
- Placebo (Placebo Comparator): Placebo (Rice Flour)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Chitin-Glucan — 3 x 500 mg capsules (tid) = 4.5 mg daily dose
  Other Names: Artinia
  Arms: High Dose Chitin-Glucan
Dietary Supplement: Low Dose Chitin-Glucan — 3 x 167 mg capsules (tid) = 1.5 g daily dose
  Other Names: Artinia
  Arms: Low Dose Chitin-Glucan
Dietary Supplement: Low Dose Chitin-Glucan + Olive Extract — 3 x 167 mg capsules (tid) = 1.5 g daily dose (C-G) + 135 mg olive extract
  Other Names: Artinia Green
  Arms: Low Dose Chitin-Glucan + Olive Extract
Dietary Supplement: Placebo — 3 x 500 mg capsules (tid)
  Other Names: Rice Flour
  Arms: Placebo

SUMMARY:
Cardiovascular diseases (CVDs), especially atherosclerotic coronary heart disease and stroke, are the leading causes of death globally. Important risk factors for CVDs include elevated serum levels of total cholesterol, low-density lipoprotein(LDL)-cholesterol, triglycerides, and low high-density lipoprotein (HDL)-cholesterol. Elevated "oxidized" LDL, a pro-inflammatory villain, has also emerged as an important risk factor for the development of CVDs. There is a growing need to identify safe and effective nutritional interventions that offer a clinical benefit aimed at reducing one more of the risk factors for CVDs. Data from many studies in humans have shown various health benefits provided by dietary fiber intake, including an inverse association with the risk of developing cardiovascular disease. The primary purpose of this study is to determine whether daily consumption for 6 weeks of chitin-glucan, a fiber purified from a microorganism, is effective at reducing the amount of oxidized LDL in humans with borderline-to-high LDL-cholesterol. The effects of chitin-glucan on other cardiovascular risk factors will also be evaluated.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVDs), especially atherosclerotic coronary heart disease and stroke, are the leading causes of death globally. Important risk factors for CVDs include elevated serum levels of total cholesterol, low-density lipoprotein (LDL)-cholesterol, triglycerides, and low high-density lipoprotein (HDL)-cholesterol levels. Oxidized LDL has also been identified as a risk factor for CVDs. There is a growing need to identify safe and effective interventions that offer a clinical benefit aimed at reducing one more of the risk factors for CVDs.

Oxidized LDL is a unique plaque-specific protein produced in the arterial wall by the oxidative modification of the apoB-100 moiety of native LDL mediated by reactive oxygen species. Oxidized LDL is a powerful atherogenic protein, which is directly involved in the initiation and progression of atherosclerosis, the main cause of coronary artery disease (CAD). It is now widely believed that for native LDL to be atherogenic, it must be converted to oxidized LDL. Oxidized LDL is found in atherosclerotic lesions and in the circulation, but not in normal arteries. Oxidized LDL is both a biomarker of accelerated atherosclerosis and a mediator of the atherosclerotic disease process. In 1998, Holvoet et al demonstrated for the first time that elevated circulating levels of oxidized LDL were found in most untreated patients with both stable CAD and acute coronary syndromes (unstable angina; acute myocardial infarction). In this landmark study, oxidized LDL levels were measured in plasma with an ELISA procedure using the oxidized LDL-specific, murine monoclonal antibody, 4E6. Mercodia's commercially available oxidized LDL ELISA kits use Holvoet's monoclonal antibody, 4E6, which is specific for oxidatively modified LDL. The 4E6 antibody is directed against a conformational epitope in the apoprotein(apo)B-100 moiety of LDL that is generated as a consequence of aldehyde substitution of the lysine residues of apoB-100.

Data from epidemiological studies have shown various health benefits provided by dietary fiber intake, including an inverse association with the risk of CVDs. As shown in several well-controlled clinical trials, various water-soluble dietary fibers reduced total cholesterol and LDL-cholesterol while HDL-cholesterol and triglycerides were not significantly influenced. Recently, the European Food Safety Authority (EFSA) authorized a health claim related to the maintenance of normal blood cholesterol concentrations for soluble cereal fibres, particularly beta-glucans from oat and barley. The beta-glucans in these cereals are non-starch polysaccharides consisting of (1→3,1→4)-beta-D-linked glucose units.

Few studies have addressed potential favorable effects of beta-glucans from micro-organisms on CVD risk factors. One clinical study examined the effects of yeast-derived beta-glucan, a glucose polymer with beta-(1→3,1→6) linkages, on serum lipids in 15 hypercholesterolemic obese men. At the end of the 8-week treatment period (15 g fiber/day in addition to the normal diet), total cholesterol levels were decreased whereas HDL-cholesterol, LDL-cholesterol and triglycerides did not differ significantly from the baseline values. A number of animal studies showed that consumption of fungi or fungal extract can lower blood cholesterol or reduce aortic atherosclerotic lesions in rabbits fed a high-cholesterol diet or in atherosclerosis-susceptible apolipoprotein E-deficient mice fed a normal. It should be noted that the fungal component(s) causing these effects have not been identified or characterized (whole mushrooms or an impure extract were tested).

Chitin-glucan is a natural component of the cell wall of microscopic fungi. Chitin-glucan can be regarded as an insoluble dietary fiber. In hamsters fed an atherogenic diet, chitin-glucan mixed with food lowered plasma triglycerides and markedly reduced the diet-induced formation of aortic fatty streak lesions. It also reduced aortic cholesterol, cardiac superoxide anion production and hepatic malondialdehyde, and increased hepatic antioxidant enzyme activities (glutathione peroxidase and superoxide dismutase). Although oxidized LDL was not measured in this study, data from an early clinical trial indicated that consumption of chitin-glucan for 28 days decreased circulating oxidized LDL by approximately 26% in healthy, normo-cholesterolemic young males.

To confirm these results in a randomized, double-blind, placebo-controlled study using males and females with broader inclusion criteria, chitin-glucan will be evaluated alone (at 1.5 and 4.5 grams per day), and in combination with olive extract (chitin-glucan at 1.5 gram per day + olive extract at 135 mg per day). There is a large body of evidence that indicates that olive oil recapitulates many of the beneficial effects on human health, including a reduced risk for developing CVDs, that are reported for intake of the Mediterranean Diet. Numerous studies performed in vitro and in vivo have concluded that polyphenolic compounds present in extra virgin olive oil play an important role in the prevention of atherosclerotic damage through their inhibition of LDL oxidation. Tyrosol and hydroxytyrosol show dose-dependent activity in this regard and are considered potent antioxidants, demonstrating activity in the micromolar range. Thus, there is a solid scientific and clinical rationale to evaluate both chitin-glucan alone and in combination with olive extract for their ability to reduce oxidized LDL.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female able to read, comprehend, and write English at sufficient level to complete study-related materials including informed consent
2. Age: 21 - 70 years
3. Body Mass Index: 18.5 - 34.9 kg/m2
4. Fasting serum LDL-cholesterol: ≥ 130 - 189.9 mg/dl
5. Willing to take supplement three times daily for 6 weeks and undergo other study-related procedures
6. Is otherwise is in general good health as determined by the principal investigator

Exclusion Criteria:

1. Known hypersensitivity or intolerance to fiber or fiber-containing products
2. Use of any investigational drugs prior to Visit 1
3. Participation in any clinical trial while participating in this trial
4. Member or family member of research staff or study sponsor involved in the conduct of this trial
5. Greater than 5% change in body weight within 1 month of Visit 1
6. Positive pregnancy test
7. Is taking lipid-altering drug therapy within four weeks prior to Visit 1. Also excluded are supplements known to have significant lipid altering effects, such as niacin (>100 mg per day), garlic (> 600 mg per day), omega-3 fatty acids (> 1 g omega-3 fatty acids per day), red yeast rice extract, phytostanols / phytosterols (> 0.5 g per day), soluble fiber (>1 g per day), chitosan (> 1 g per day) and conjugated linoleic acid (CLA; > 3 g per day)
8. Excluded concurrent medications are: systemic corticosteroids (nasal and inhaled corticosteroids are permitted), orlistat, bile acid resins, no more than 1 g of prescription omega-3 fatty acids, cyclical or non-continuous hormone therapy (estrogen or testosterone)
9. No more than 2 units of ethanol per day. Units are defined as 1.5 ounces of 80 proof alcohol per day, e.g. 2 twelve ounce cans of beer per day.
10. Has a fasting serum triglyceride > 300 mg/dl
11. Has a diagnosis of type 1 or type 2 diabetes mellitus or fasting glucose > 126 mg/dl
12. Has a serum thyroid-stimulating hormone (TSH) higher than 1.5 times the upper limit of normal for the laboratory
13. Is breast feeding, pregnant, or planning on becoming pregnant during the duration of the study
14. Known cardiovascular disease or stroke, except for conditions that are deemed clinically insignificant by Principle Investigator or Sub-investigator, or study site physician (e.g. clinically insignificant atherosclerotic lesions observed by imaging studies).
15. History of significant gastrointestinal disease such as severe constipation, diarrhea, malabsorptive disease, inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis)
16. History of severe psychiatric illness which in the opinion of the investigator would interfere with the optimal participation in the study
17. History if cancer within 5 years of Visit 1 (except for successfully treated basal and squamous cell carcinoma of the skin)
18. Known human immunodeficiency virus (HIV) seropositivity
19. History of bariatric surgery
20. Aspartate aminotransferase (AST) or alanine transaminase (ALT) > 3 times the upper limit of normal
21. Creatine kinase (CK) ≥ 3 times the upper limit of normal, unless explained by recent physical activity or trauma; or > 5 times the upper limit of normal, irrespective of circumstance
22. Creatinine ≥ 1.5 mg/dl
23. Individuals who in the opinion of the principal investigator have a risk of non-compliance to the study procedures or who are otherwise not appropriate to include in this clinical trail

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Oxidized LDL | After 4 and 6 weeks

SECONDARY OUTCOMES:
Total cholesterol | After 4 and 6 weeks
LDL-cholesterol | After 4 and 6 weeks
HDL-cholesterol | After 4 and 6 weeks
Triglycerides | After 4 and 6 weeks
Glucose | After 4 and 6 weeks
Insulin | After 4 and 6 weeks
F2-isoprostanes (urine) | After 4 and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph L Evans, PhD, Study Director — Stratum Nutrition; James Anderson, MD, Study Chair — Consultant / Advisor (Stratum and KitoZyme); Ray Cooper, PhD, Study Director — Stratum Nutrition; Veronique Maquet, PhD, Study Director — Kitozyme
Locations (3):
- United States (2):
  - Provident Clinical Research and Consulting, Addison, Illinois
  - Louisville Metabolic and Atherosclerosis Research Center (L-MARC), Louisville, Kentucky
- KGK Synergize, London, Ontario, Canada

REFERENCES:
- [Background] Berecochea-Lopez A, Decorde K, Ventura E, Godard M, Bornet A, Teissedre PL, Cristol JP, Rouanet JM. Fungal chitin-glucan from Aspergillus niger efficiently reduces aortic fatty streak accumulation in the high-fat fed hamster, an animal model of nutritionally induced atherosclerosis. J Agric Food Chem. 2009 Feb 11;57(3):1093-8. doi: 10.1021/jf803063v. PMID 19154104
- [Background] Jonker D, Kuper CF, Maquet V, Nollevaux G, Gautier S. Subchronic (13-week) oral toxicity study in rats with fungal chitin-glucan from Aspergillus niger. Food Chem Toxicol. 2010 Oct;48(10):2695-701. doi: 10.1016/j.fct.2010.06.042. Epub 2010 Jun 30. PMID 20600523
- [Background] Anderson JW, Baird P, Davis RH Jr, Ferreri S, Knudtson M, Koraym A, Waters V, Williams CL. Health benefits of dietary fiber. Nutr Rev. 2009 Apr;67(4):188-205. doi: 10.1111/j.1753-4887.2009.00189.x. PMID 19335713
- [Background] Huang H, Mai W, Liu D, Hao Y, Tao J, Dong Y. The oxidation ratio of LDL: a predictor for coronary artery disease. Dis Markers. 2008;24(6):341-9. doi: 10.1155/2008/371314. PMID 18688083
- [Background] Neyrinck AM, Possemiers S, Verstraete W, De Backer F, Cani PD, Delzenne NM. Dietary modulation of clostridial cluster XIVa gut bacteria (Roseburia spp.) by chitin-glucan fiber improves host metabolic alterations induced by high-fat diet in mice. J Nutr Biochem. 2012 Jan;23(1):51-9. doi: 10.1016/j.jnutbio.2010.10.008. Epub 2011 Mar 15. PMID 21411304
- [Result] Bays HE, Evans JL, Maki KC, Evans M, Maquet V, Cooper R, Anderson JW. Chitin-glucan fiber effects on oxidized low-density lipoprotein: a randomized controlled trial. Eur J Clin Nutr. 2013 Jan;67(1):2-7. doi: 10.1038/ejcn.2012.121. Epub 2012 Sep 5. PMID 22948945
- See also: KitoZyme — http://www.kitozyme.com
- See also: Provident Clinical Research and Consulting — http://www.providentcrc.com/